CLINICAL TRIAL: NCT06573593
Title: Efficacy and Safety of JAK Inhibitors in Patients With Alopecia Areata: a Single-center, Real-world Study
Brief Title: Efficacy and Safety of JAK Inhibitors in Patients With AA: RWE Study
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 20240699
Record Dates: First submitted 2024-08-25; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-07

CONDITIONS: Alopecia Areata; Janus Kinase Inhibitors
MeSH Terms: conditions — Alopecia Areata | interventions — tofacitinib; baricitinib; ruxolitinib; upadacitinib; abrocitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Tofacitinib treated group: In the real-world settings, patients with AA treated with tofacitinib.
  Interventions: Drug: Tofacitinib
- Baritinib treated group: In the real-world settings, patients with AA treated with baritinib.
  Interventions: Drug: Baricitinib
- Ruxolitinib treated group: In the real-world settings, patients with AA treated with ruxolitinib
  Interventions: Drug: Ruxolitinib
- Upadacitinib treated group: In the real-world settings, patients with AA treated with upadacitinib.
  Interventions: Drug: Upadacitinib
- Abrocitinib treated group: In the real-world settings, patients with AA treated with abhicitinib.
  Interventions: Drug: Abrocitinib
- Ritlecitinib treated group: In the real-world settings, patients with AA treated with ritlecitinib.
  Interventions: Drug: Ritlecitinib

INTERVENTIONS:
Drug: Tofacitinib — In the real-world settings, patients with AA treated with tofacitinib.
  Groups: Tofacitinib treated group
Drug: Baricitinib — In the real-world settings, patients with AA treated with Baricitinib.
  Groups: Baritinib treated group
Drug: Ruxolitinib — In the real-world settings, patients with AA treated with Ruxolitinib.
  Groups: Ruxolitinib treated group
Drug: Upadacitinib — In the real-world settings, patients with AA treated with Upadacitinib.
  Groups: Upadacitinib treated group
Drug: Abrocitinib — In the real-world settings, patients with AA treated with Abrocitinib.
  Groups: Abrocitinib treated group
Drug: Ritlecitinib — In the real-world settings, patients with AA treated with Ritlecitinib.
  Groups: Ritlecitinib treated group

SUMMARY:
The introduction of Janus Kinase inhibitors (JAKi) seems to revolutionize the field of alopecia areata (AA) therapeutics. However, the ideal JAKi is not yet settled and the real-world data are still missing. To provide evidence about effectiveness and safety of different JAKi including tofacitinib, baricitinib, ritlecitinib，abrocitinib, upadacitinib and ifidancitinib in real-world settings and describe baseline disease characteristics and patients profiles that are considered good candidates for JAKi in the daily practice. Furthermore, we intended to investigate the efficacy and safety of JAK Inhibitors in patients With AA, as well as to provide clinical evidence for the clinicians and patients when they formulate individualized treatment plans.

ELIGIBILITY:
Inclusion Criteria:

* Patients with alopecia areata between 2 to 18 years old
* Patients diagnosed with alopecia areata according to AA guideline
* AA Patients treated with JAKi including tofacitinib, baricitinib, ritlecitinib，abrocitinib, upadacitinib and ifidancitinib for more than 3 months

Exclusion Criteria:

* Patients had previously received hair implants
* Other alopecia
* Other diseases may induce alopecia including psoriasis, lichen planus, et al.
* Unable to estimate SALT score at baseline or at follow-up
* Patients are participating in other clinical trials

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with alopecia areata treated with JAKi including tofacitinib, baricitinib, ritlecitinib，abrocitinib, upadacitinib and ifidancitinib for more than 3 months in Department of Dermatology, Second Affiliated Hospital, Zhejiang University School of Medicine
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean SALT | at week 24
  Reduction of Severity of Alopecia Tool (SALT) score compared with baseline
SALT50 | at week 24
  Percentage of patient with more than 50% improvement in SALT score
SALT75 | at week 24
  Percentage of patient with more than 70% improvement in SALT score

SECONDARY OUTCOMES:
Mean SALT | at week 12, 36, 48, 56
  Reduction of Severity of Alopecia Tool (SALT) score compared with baseline
SALT50 | at week 12, 36, 48, 56
  Percentage of patient with more than 75% improvement in SALT score
SALT75 | at week 12, 36, 48, 56
  Percentage of patient with more than 50% improvement in SALT score
Safety profile | at week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56
  Any adverse events including infection, hypohepatia, thrombus, gastrointestinal reaction and any other system events.

CONTACTS AND LOCATIONS:
Overall Officials: Xianjie Wu, Ph.D, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No